CLINICAL TRIAL: NCT03550612
Title: Neonatal Hypoxic Ischemic Encephalopathy:Targeting Early Diagnosis and Management of Associated Comorbidities
Brief Title: Neonatal Hypoxic Ischemic Encephalopathy:Early Diagnosis and Management of Comorbidities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ASAli, Principle investigator, Assiut University
Other Study IDs: NHIE
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Neonatal Hypoxic Ischemic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates with hypoxic ischemic encephalopathy: Cranial ultrasound,Magnetic resonant imaging and amplitude integrated encephalogram performed to All neonates with hypoxic ischemic encephalopathy in period between January 2010 to December 2015.
  Interventions: Diagnostic Test: magnetic resonant imaging,cranial ultrasound.; Diagnostic Test: Amplitude integrated electroencephalogram

INTERVENTIONS:
Diagnostic Test: magnetic resonant imaging,cranial ultrasound. — Magnetic resonant image performed at term gestation neonate suffer of hypoxic ischemic encephalopathy and its results will be analysed in details and classified according to global score of magnetic resonant image injury.Cranial ultrasound results will be analysed regards (periventricular - interventricular haemorrhage-Ventricular size-basal ganglia, thalamus and cerebellum affection) and Doppler (peak systolic flow velocity-end diastolic peak flow velocity-mean velocity and resistance index).Cerebral bleeding will be diagnosed be cranial ultrasound and confirmed be standard magnetic resonant image in term equivalent age.
Diagnostic Test: Amplitude integrated electroencephalogram — Amplitude integrated electroencephalogram before and during cooling will be assessed and classified according to Hellstrom Westas et al 2006 and it will be compared with the results of cranial ultrasound and magnetic resonant imaging.
  Neurodevelopment study at 12 and 14 month age using Bayley ɪɪɪ score will be compared with the results of cranial ultrasound,magnetic resonant imaging and Amplitude integrated electroencephalogram.

SUMMARY:
Perinatal asphyxia is common cause of acquired neonatal brain injury in neonates associated with hypoxic-ischemic encephalopathy, leading to long-term neurologic complication or death. In 2000, the neonatal mortality rate in Egypt was found to be 25 per 1000 live birth. In this survey, hypoxic ischemic encephalopathy accounts for 18% of neonatal mortality and is the second most common cause of neonatal death.

DETAILED DESCRIPTION:
Cerebral palsy as complication of hypoxic ischemic encephalopathy is common problem in Egypt.cerebral palsy is associated with many problems (cognitive disability-epilepsy-visual and hearing problems) that make great economic burden on their family and health care system. In 2010, the prevalence of cerebral palsy in El-Kharga District new valley described 2.04 cases of cerebral palsy every 1000 child.hypoxic ischemic encephalopathy was the second most common cause of cerebral palsy with prematurity the most common. 70.5% of children with cerebral palsy had severe mental retardation and 52% suffer from active epilepsy. An observational study on 224 cerebral palsy case from Tanta University found that 80.8% of patients with cerebral palsy had cognitive disorder, 36% had epilepsy, 25% loss of vision and 16% hearing problems. This health conditions provide a significant financial burden on the health system in Egypt.

There are two problems regard dealing with cases of hypoxic ischemic encephalopathy in Egypt, First one is early diagnosis and second is description of its severity. Assessment of the severity of cerebral injury and neurological outcome in infants with hypoxic ischemic encephalopathy is important for prognosis and stratifying the clinical management. Neurophysiological tests, including amplitude-integrated electroencephalogram , biochemical markers, and neuroimaging like (Trans cranial ultrasound - Magnetic resonance imaging) have been used to assess prognosis and predict long-term outcome. In our neonatal unit investigators perform routine cranial ultrasound to all cases of hypoxic ischemic encephalopathy.Cranial ultrasound is cheap, available, and easily performed bedside examination. However cranial ultrasound is limited in specificity and sensitivity in diagnosis of Hypoxic ischemic encephalopathy and prediction of prognosis.

Magnetic resonant imaging might provide the best information on structural brain lesions associated with long-term neurological impairment but is not available for immediate diagnostics on neonatal unit. Amplitude integrated electroencephalography is unfortunately not routinely performed in Egyptian neonatal units. It might improve early detection of Hypoxic ischemic encephalopathy and risk stratification accordingly.

Cerebral bleeding and infection are commonly described comorbidities in Hypoxic ischemic encephalopathy associated with the poor prognosis. Coagulopathy is common problem in asphyxiated infants. It is associated with asphyxia and therapeutic hypothermia (standardized treatment of hypoxia). Coagulopathy can cause bleeding in serious organs like brain that make the prognosis of Hypoxia bad and control of seizure difficult.

ELIGIBILITY:
Inclusion Criteria:

* >36 weeks gestational age babies undergoes therapeutic hypothermia within 6 hours after birth after fulfilling the cooling criteria:
* Apgar score ≤ 5 at 10 minutes after birth.
* Need resuscitation 10 minutes after birth.
* Acidosis PH≤7 at 60 minutes.
* Base deficit ≥16 mmoL ∕ L at 60 minutes.

Exclusion Criteria:

* Birth weight ≤1.8kg.
* Congenital and genetic conditions affect neurodevelopment.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all neonates with hypoxic ischemic encephalopathy treated by therapeutic hypothermia 6 hours after birth in period between January 2010 to December 2015.One hundred cases will be included in the study as fifteen to twenty case of HIE admitted for therapeutic hypothermia treatment at the hospital every year.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Compare results of cranial ultrasound with Magnetic resonant imaging to improve quality of cranial ultrasound to early diagnosis of hypoxic ischemic encephalopathy | 3 weeks age.
  Cranial ultrasound results will be analysed regards (periventricular - interventricular haemorrhage-Ventricular size-basal ganglia, thalamus and cerebellum affection) and Doppler (peak systolic flow velocity-end diastolic peak flow velocity-mean velocity and resistance index).magnetic resonant imaging performed at term gestation results will be analysed in details and classified according to global score of magnetic resonant imaging injury (mild, moderate and severe injury) and compare it with results of cranial ultrasound

SECONDARY OUTCOMES:
Detect incidence of intracranial haemorrhage in asphyxiated newborn treated by therapeutic hypothermia. | 12 month
  Analysis of perinatal risk factors associated with increase incidence of intracranial hemorrhage.and coagulation limits after that intracranial haemorrhage occurs and transfusion limits decrease incidence of intracranial haemorrhage.
Detection of associated infection in asphyxiated newborn treated by therapeutic hypothermia. | 1 month
  Detection of associated infection that increase seizure activity and make it difficult to control.C-reactive protein and blood culture will be the gold standard to diagnosis associated infection, suspicious sepsis on C-reactive protein ≥ 10 and confirmed by blood culture.
Ability of cranial ultrasound in early diagnosis of intracranial haemorrhage. | 1 month age
  By compare results of cranial ultrasound with standard magnetic resonant imaging
Compare results of diagnostic methods of hypoxic ischemic encephalopathy with neurodevelopmental study of the baby at 12 month | 12 month age
  Compare results of magnetic resonant imaging,Cranial ultrasound and amplitude integrated encephalogram in babies with Hypoxic ischemic encephalopathy undergoes therapeutic cooling with neurodevelopmental score at 12 month age.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pierrat V, Haouari N, Liska A, Thomas D, Subtil D, Truffert P; Groupe d'Etudes en Epidemiologie Perinatale. Prevalence, causes, and outcome at 2 years of age of newborn encephalopathy: population based study. Arch Dis Child Fetal Neonatal Ed. 2005 May;90(3):F257-61. doi: 10.1136/adc.2003.047985. PMID 15846019
- [Background] Campbell O, Gipson R, el-Mohandes A, Issa AH, Matta N, Mansour E, Mohsen L. The Egypt National Perinatal/Neonatal Mortality Study 2000. J Perinatol. 2004 May;24(5):284-9. doi: 10.1038/sj.jp.7211084. PMID 15042109
- [Background] El-Tallawy HN, Farghaly WM, Shehata GA, Metwally NA, Rageh TA, Abo-Elfetoh N. Epidemiology of cerebral palsy in El-Kharga District-New Valley (Egypt). Brain Dev. 2011 May;33(5):406-11. doi: 10.1016/j.braindev.2010.07.011. Epub 2010 Aug 24. PMID 20797827
- [Background] Merchant N, Azzopardi D. Early predictors of outcome in infants treated with hypothermia for hypoxic-ischaemic encephalopathy. Dev Med Child Neurol. 2015 Apr;57 Suppl 3:8-16. doi: 10.1111/dmcn.12726. PMID 25800487
- [Background] Forman KR, Diab Y, Wong EC, Baumgart S, Luban NL, Massaro AN. Coagulopathy in newborns with hypoxic ischemic encephalopathy (HIE) treated with therapeutic hypothermia: a retrospective case-control study. BMC Pediatr. 2014 Nov 3;14:277. doi: 10.1186/1471-2431-14-277. PMID 25367591
- [Background] Bednarek N, Mathur A, Inder T, Wilkinson J, Neil J, Shimony J. Impact of therapeutic hypothermia on MRI diffusion changes in neonatal encephalopathy. Neurology. 2012 May 1;78(18):1420-7. doi: 10.1212/WNL.0b013e318253d589. Epub 2012 Apr 18. PMID 22517107
- [Background] Tao JD, Mathur AM. Using amplitude-integrated EEG in neonatal intensive care. J Perinatol. 2010 Oct;30 Suppl:S73-81. doi: 10.1038/jp.2010.93. PMID 20877412